CLINICAL TRIAL: NCT05546125
Title: A Non-interventional Study to Further Characterize the Safety and Effectiveness of Sildenafil in the Treatment of Pulmonary Arterial Hypertension (PAH) in Adults From China in a Real World Setting
Brief Title: a Non-interventional Study of Sildenafil in the Treatment of Pulmonary Arterial Hypertension (PAH) in Adults From China
Status: Completed | Type: Observational
Sponsor: Pfizer Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Other Study IDs: A1481336
Record Dates: First submitted 2022-08-30; First posted 2022-09-19 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Pulmonary Arterial Hypertension (PAH)
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: as per Physician's prescription — Participants need to take the Revatio as per Physician's prescription

SUMMARY:
This observational study will involve analysis of data collected by the National Rare Disease Registry or medical records .The study will describe outcomes only in PAH(Pulmonary arterial hypertension) patients treated with sildenafil; there will be no comparison with another treatment group.

Approximately 100 adults with PAH will be recruited in China hospitals This NIS(non-interventional study) data will be recorded by a physician in the medical records, during the patients' clinical visits, and in the electronic Case Report Forms (CRF).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at study index date; (The index date (i.e., Day 1 of the study) is the date when the first sildenafil dose was actually taken, after Revatio® is approved by China authority)
* A diagnosis of PAH with a mean pulmonary artery pressure of ≥25 mmHg and a mean pulmonary capillary wedge pressure of ≤15 mmHg by right heart catheterization;
* Initiated sildenafil for the treatment of their PAH based on treatment suggestion from physician ;(Patients who have received sildenafil or are receiving sildenafil are eligible to participate in this study if they met the above inclusion criteria and were ready to start sildenafil (Revatio®) for treatment at screening;)
* Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

* No

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will comprise patients with PAH (including idiopathic pulmonary arterial hypertension, PAH associated with connective tissue disease, and PAH associated with congenital heart disease patients) Patients must meet all of the inclusion criterias to be eligible for inclusion in this study
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-12-23 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent Adverse Events (TEAEs) | From baseline to week24
  Incidence of TEAEs and the type of TEAEs
Serious adverse events (SAEs) | From baseline to week24
  Incidence of SAE and the type of SAE

SECONDARY OUTCOMES:
6-MWD (6-minute walk distance) | baseline, week 12, week24
  Change in 6-minute walk distance (6-MWD)

CONTACTS AND LOCATIONS:
Locations (7):
- China (7):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital, Guangdong, Guangzhou
  - The Second Xiangya Hospital Of Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Affiliated Hospital of Jining Medical College, Jining, Shandong
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Yanan Hospital of Kunming City, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No